CLINICAL TRIAL: NCT00793962
Title: A Phase Ⅲ Randomized Clinical Trial of Postmastectomy Hypofractionation Radiotherapy in High-risk Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shu lian Wang, M.D., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2008A06
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; mastectomy; radiotherapy; fractionation
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypofractionation radiotherapy (Experimental): breast cancer women with mastectomy high-risk: T3-4 and/or 4 or more axillary nodes involvement postmastectomy hypofractionation radiotherapy of 43.5Gy/15f/3w to the chest wall and supraclavicular nodal region
  Interventions: Radiation: hypofractionation radiotherapy
- conventional fractionation radiotherapy (Active Comparator): breast cancer women with mastectomy high-risk with T3-4 and/or 4 or more axillary nodes postmastectomy conventional fractionation radiotherapy of 50Gy/25f/5w to the chest wall and supraclavicular nodal region
  Interventions: Radiation: conventional fractionation radiotherapy

INTERVENTIONS:
Radiation: hypofractionation radiotherapy — radiotherapy of 43.5Gy/15f/3w to the chest wall and supraclavicular nodal region
  Other Names: radiotherapy
  Arms: hypofractionation radiotherapy
Radiation: conventional fractionation radiotherapy — 50Gy/25/f/5w
  Other Names: radiotherapy
  Arms: conventional fractionation radiotherapy

SUMMARY:
The purpose of this study is to compare the efficacy and toxicities of hypofractionation radiotherapy with conventional fractionation radiotherapy in breast cancer patients treated with mastectomy.It is hypothesized that the efficacy and toxicities are similar between the two groups.

DETAILED DESCRIPTION:
Eligible breast cancer patients with mastectomy and axillary dissection are randomized into 2 groups:conventional fractionation radiotherapy of 50 Gy in 25 fractions within 5 weeks to ipsilateral chest wall and supraclavicular nodal region,and hypofractionation radiotherapy of 43.5Gy in 15 fractions within 3 weeks to the same region.

During and after radiotherapy, the patients are followed and the efficacy and toxicities of radiotherapy are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Ipsilateral histologically confirmed invasive breast cancer
* Undergone total mastectomy and axillary dissection
* T3-4,or >=4 positive axillary lymph nodes
* Fit for chemotherapy(if indicated),endocrine therapy(if indicated)and postoperative irradiation
* Written,informed consent
* cT3-4,or cN2, or pathological positive axillary lymph nodes during mastectomy for patients who had received neoadjuvant chemotherapy or hormone therapy
* no supraclavicular or internal mammary nodes metastases
* no distant metastases
* enrollment date no more than 8 months after surgery or no more than 2 months after chemotherapy for patients who didn't receive neoadjuvant systemic therapy.
* enrollment date no more than 2 months after surgery for patients who had received neoadjuvant systemic therapy and didn't need adjuvant chemotherapy.

Exclusion Criteria:

* Patients who undergone previous irradiation to the ipsilateral chest wall and supraclavicular region
* Previous or concurrent malignant other than non-melanomatous skin cancer
* Unable or unwilling to give informed consent
* bilateral breast cancer
* immediate or delayed ipsilateral breast cancer reconstruction

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2008-06; Primary Completion 2016-05 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
locoregional control rate | 5 years
  ipsilateral chest wall, axilla, supraclavicular and internal mammary nodal relapse

SECONDARY OUTCOMES:
overall survival | 5 years
  any death

CONTACTS AND LOCATIONS:
Overall Officials: shu-lian wang, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Ye-xiong Li, M.D., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Yang J, Qi SN, Fang H, Song YW, Jin J, Liu YP, Wang WH, Yang Y, Tang Y, Ren H, Chen B, Lu NN, Tang Y, Li N, Jing H, Wang SL, Li YX. Cost-effectiveness of postmastectomy hypofractionated radiation therapy vs conventional fractionated radiation therapy for high-risk breast cancer. Breast. 2021 Aug;58:72-79. doi: 10.1016/j.breast.2021.04.002. Epub 2021 Apr 19. PMID 33933925
- [Derived] Wang SL, Fang H, Song YW, Wang WH, Hu C, Liu YP, Jin J, Liu XF, Yu ZH, Ren H, Li N, Lu NN, Tang Y, Tang Y, Qi SN, Sun GY, Peng R, Li S, Chen B, Yang Y, Li YX. Hypofractionated versus conventional fractionated postmastectomy radiotherapy for patients with high-risk breast cancer: a randomised, non-inferiority, open-label, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):352-360. doi: 10.1016/S1470-2045(18)30813-1. Epub 2019 Jan 30. PMID 30711522